CLINICAL TRIAL: NCT04936308
Title: A Phase 3B, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Participants With Active Psoriatic Arthritis Who Had an Inadequate Response and/or Intolerance to One Prior Anti-Tumor Necrosis Factor Alpha Agent
Brief Title: Guselkumab in Active Psoriatic Arthritis Participants With Inadequate Response/Intolerance to One Prior Anti-TNF Alpha Agent
Acronym: SOLSTICE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109039; CNTO1959PSA3005 (Other: Janssen Research & Development, LLC); 2021-000482-32 (EudraCT Number); 2023-504715-33-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab and Placebo (Experimental): Participants will receive guselkumab and placebo subcutaneously (SC) to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab SC.
  Interventions: Drug: Guselkumab
- Group 3: Placebo Followed by Guselkumab (Experimental): Participants will receive placebo SC and will cross over to receive guselkumab SC.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive guselkumab as SC injection.
  Other Names: Tremfya; CNTO1959
Drug: Placebo — Participants will receive matching placebo as SC injection.
  Arms: Group 1: Guselkumab and Placebo; Group 3: Placebo Followed by Guselkumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab treatment in participants with active psoriatic arthritis (PsA) and inadequate response (IR) and/or intolerance to a prior anti-tumor necrosis factor (TNF) by assessing the reduction in signs and symptoms of PsA.

DETAILED DESCRIPTION:
PsA is a chronic, immune-mediated inflammatory disease characterized by peripheral joint inflammation, enthesitis, dactylitis, axial disease, and the skin lesions associated with psoriasis. Guselkumab is a fully human monoclonal antibody (mAb) that binds to p19 protein subunit of interleukin (IL)-23 and blocks the binding of extracellular IL-23 to the cell surface IL-23 receptor, inhibiting IL-23 specific intracellular signaling, subsequent activation, and cytokine production. The primary hypothesis of this study is that guselkumab is superior to placebo as assessed by the proportion of participants who had an inadequate response (IR) and/or intolerance to one prior anti-tumor necrosis factor (anti-TNF) achieving an American College of Rheumatology 20 (ACR 20) response at Week 24. This study will consist of a screening phase (up to 6 weeks), blinded treatment phase (approximately up to 2 years), which includes a placebo-controlled period from Week 0 to Week 24, and an active-controlled treatment phase from Week 24 to Week 100, and safety follow-up phase (Week 112). Safety assessments will include physical examinations, vital signs, height, weight, electrocardiograms, and clinical safety laboratory assessments. The total duration of the study will be up to 118 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of active psoriatic arthritis (PsA) for at least 6 months before the first administration of study agent and meet Classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: at least 3 swollen joints and at least 3 tender joints at screening and at baseline; and C-reactive protein (CRP) greater than or equal to (>=) 0.3 milligrams per deciliter (mg/dL) at screening from the central laboratory
* Have at least one of the following PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis, with at least one psoriatic plaque of >= 2 centimeters (cm) diameter and/or nail changes consistent with psoriasis, or documented history of plaque psoriasis
* Have an inadequate response and/or intolerance to anti-tumor necrosis factor alpha (TNF alpha) therapy, defined as presence of active PsA despite previous treatment with one prior anti-TNF alpha agent

Exclusion Criteria:

* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy in the treatment of PsA, including but not limited to rheumatoid arthritis, ankylosing spondylitis/nonradiographic axial spondyloarthritis, systemic lupus erythematosus, or Lyme disease
* Has received more than 1 prior anti-tumor necrosis factor (TNF) alpha agent (or biosimilars)
* Has ever received Janus kinase (JAK) inhibitor including but not limited to tofacitinib, baricitinib, filgotinib, peficitinib, decernotinib, upadacitinib or any other investigational JAK inhibitor
* Has received any systemic immunosuppressants (example, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study intervention
* Has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients
* Has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection (example, bronchiectasis), recurrent urinary tract infection (example, recurrent pyelonephritis or chronic non-remitting cystitis), fungal infection (example, mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2026-07-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (169):
- United States (50):
  - Arthritis Associates, Mountain Brook, Alabama
  - Arizona Arthritis and Rheumatology Research PLLC, Avondale, Arizona
  - Arizona Arthritis and Rheumatology Research PLLC, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Research PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research PLLC, Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Associates, Sun City, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - Unity Health-White County Medical Center, Searcy, Arkansas
  - Newport Huntington Medical Group, Huntington Beach, California
  - Medvin Clinical Research, Thousand Oaks, California
  - Medvin Clinical Research, Tujunga, California
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Omega Research Consultants, DeBary, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Clinic of Robert Hozman, Skokie, Illinois
  - The Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Klein And Associates M D P A, Hagerstown, Maryland
  - Great Lakes Center of Rheumatology, Lansing, Michigan
  - Arthritis and Rheumatology Center of MI, Okemos, Michigan
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - St. Paul Rheumatology P A, Eagan, Minnesota
  - Arthritis Consultants, St Louis, Missouri
  - Arthritis Rheumatic And Back Disease Associates, Voorhees Township, New Jersey
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Arthritis and Osteoperosis Associates of New Mexico, Las Cruces, New Mexico
  - Buffalo Rheumatology and Medicine PLLC, Orchard Park, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - STAT Research, Inc., Vandalia, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Rheumatology Associates of Oklahoma, Oklahoma City, Oklahoma
  - Dr. Ramesh Gupta, Memphis, Tennessee
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Adriana Pop Moody MD Clinic PA, Corpus Christi, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Precision Comprehensive Clinical Research Solutions, Fort Worth, Texas
  - West Texas Clinical Research, Lubbock, Texas
  - Southwest Rheumatology Research LLC, Mesquite, Texas
  - Texas Rheumatology Care, Plano, Texas
  - Advanced Rheumatology of Houston, The Woodlands, Texas
  - DM Clinical Research, Tomball, Texas
  - Arthritis And Osteoporosis Clinic, Waco, Texas
  - Arthritis Northwest PLLC, Spokane, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (7):
  - Cosultorios Reumatologógicos Pampa, Buenos Aires
  - OMI, Buenos Aires
  - CIPREC, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Hospital Central Militar Cirujano Mayor Dr Cosme Argerich, Buenos Aires
  - Instituto de Reumatología Mendoza, Mendoza
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Australia (4):
  - Southern Clinical Research, Hobart
  - Liverpool Hospital, Liverpool
  - Skin Health Institute Inc., Melbourne
  - Eastern Health - Box Hill Hospital, Melbourne
- Bulgaria (9):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Medical Center Unimed Plovdiv, Plovdiv
  - UMHAT Kaspela, Plovdiv
  - Diagnosis-consulting centre-1, Rousse
  - Military Medical Academy, Sofia
  - UMHAT St. Ivan Rilski, Sofia
  - ASIMP Rheumatology Centre St Irina EOOD, Sofia
  - University Multiprofile Hospital Sofiamed Sofia, Sofia
  - Medical Centre Synexus, Sofia
- Czechia (7):
  - RHEUMA s r o, Břeclav
  - L K N Arthrocentrum, Hlučín
  - MUDr Rosypalova s r o, Ostrava
  - Arthrohelp S.R.O., Pardubice
  - Revmatologicky ustav, Prague
  - Medical Plus S R O, Uherské Hradiště
  - PV Medical S R O, Zlín
- Hungary (8):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Uno Medical Trials Ltd., Budapest
  - Debreceni Egyetem, Kenézy Gyula Egyetemi Oktatókórház, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szegedi Tudományegyetem, ÁOK, Szent-Györgyi Albert Klinikai Központ, Szeged
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Malaysia (4):
  - Hospital Selayang, Batu Caves
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Tuanku Jaafar, Seremban
- Poland (16):
  - Nzoz Bif Med, Bytom
  - Centrum Kliniczno Badawcze, Elblag
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Medyczne Promed, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Twoja Przychodnia PCM, Poznan
  - Centrum Medyczne, Poznan
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Rheuma Medicus Sp z o o, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Puerto Rico (3):
  - GCM Medical Group, San Juan
  - Mindful Medical Research, San Juan
  - FDI Clinical Research, San Juan
- Russia (20):
  - Altay Medical State University, Barnaul
  - Chelyabinck Regional Clinical Hospital, Chelyabinsk
  - Chelyabinsk Regional Clinical Dermatovenerological Dispensary, Chelyabinsk
  - Kemerovo State Medical University, Kemerovo
  - LLL Medical Center Revma-Med, Kemerovo
  - LLC Family Outpatient Clinic # 4, Korolyov
  - Krasnodar Clinical Dermatovenerologic Dispensary, Krasnodar
  - Regional SBI of PH Krasnoyarsk Regional Clinical hospital #20 named after I.S. Berzon, Krasnoyarsk
  - Clinical-Diagnostic Center Euromedservice, JSC, Moscow
  - FGBU Research Institute of Rheumatology named V.A.Nasonova, Moscow
  - GBUZ of Moscow Region 'Moscow Region SRI n.a. Vladimirskyi', Moscow
  - GBOU VPO Orenburg State Medical University, Orenburg
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - St. Petersburg GBUZ Clinical Reumatological Hospital 25, Saint Petersburg
  - X7 Clinical Research Company Limited, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Smolensk regional hospital on Smolensk railway station, Smolensk
  - GBUZ of Samara Region 'Tolyatti City Clinical Hospital 5', Tolyatti
  - Tula Regional Clinical Dermatovenerological Dispensary, Tula
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
- Spain (7):
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Quiron Madrid Pozuelo, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Clinica Gaias, Santiago de Compostela
  - Hosp. Quiron Sagrado Corazon, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Turkey (Türkiye) (14):
  - Adana City Hospital, Adana
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Uludag University Medical Faculty, Bursa
  - Pamukkale University Medical Faculty, Denizli
  - Osmangazi University Medical Faculty, Eskişehir
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Kartal Dr Lutfi Kirdar sehir Hastanesi, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- Ukraine (15):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Municipal non-commercial enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - City Clinical Hospital No. 2, Kryvyi Rih
  - Medical Center LLC 'Harmony of Beauty', Kyiv
  - Medical Center of 'Institute of Rheumatology', LLC, Kyiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - LLC Medical House, Odesa
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - Vinnitsia Regional Clinical Hospital n.a. M. I. Pyrogov, Vinnytsia
  - Medical Center LLC 'Modern Clinic', Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Ogdie A, Merola JF, Mease PJ, Ritchlin CT, Scher JU, Lafferty KP, Chan D, Chakravarty SD, Langholff W, Wang Y, Choi O, Krol Y, Gottlieb AB. Efficacy and safety of guselkumab in patients with active psoriatic arthritis who had inadequate efficacy and/or intolerance to one prior tumor necrosis factor inhibitor: study protocol for SOLSTICE, a phase 3B, multicenter, randomized, double-blind, placebo-controlled study. BMC Rheumatol. 2024 May 21;8(1):20. doi: 10.1186/s41927-024-00386-7. PMID 38773563

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Followed by Guselkumab 100 mg: Participants received placebo matched to guselkumab subcutaneous (SC) injections every 4 weeks (q4w) from Week 0 through Week 20. At Week 24, participants crossed over to receive guselkumab 100 mg SC injections q4w from Week 24 through Week 100.
- Guselkumab 100 mg q8w: Participants received guselkumab 100 mg SC injections at Weeks 0 and 4, then every 8 weeks (q8w) from Week 12 to Week 100 and placebo matched to guselkumab SC injections at Week 8 then q8w through Week 96 to maintain the blind.
- Guselkumab 100 mg q4w: Participants received guselkumab 100 mg SC injections q4w from Week 0 through Week 100.
Period: Overall Study
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 150 | 152 (Includes 1 participant that was randomized and treated at 2 sites simultaneously and was excluded from all analysis sets.) | 151 (Includes 1 participant that was randomized and treated at 2 sites simultaneously and was excluded from all analysis sets.)
Full Analysis Set (All participants who were randomized in the study. This excludes the 1 participant that was randomized and treated twice.) | 150 | 151 | 150
Completed | 138 | 144 | 141
Not Completed | 12 | 8 | 10
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 0
Not completed — Excluded from analysis (Enrolled and dosed at 2 sites) | 0 | 1 | 1
Not completed — Completed protocol-required follow-up | 1 | 2 | 2
Not completed — Discontinued study intervention and were being followed | 2 | 2 | 4
Not completed — Other | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized in the study and included in the analyses.
Groups:
- Placebo: Participants received placebo matched to guselkumab subcutaneous (SC) injections every 4 weeks (q4w) from Week 0 through Week 20. At Week 24, participants crossed over to receive guselkumab 100 mg sc injections every 4 weeks from Week 24 through Week 100.
- Guselkumab 100 mg q4w: Participants received guselkumab 100 mg subcutaneous injections every 4 weeks from Week 0 through to end of study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w | Total
Number analyzed (Participants) | 150 | 151 | 150 | 451
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (12.59) | 51.9 (12.91) | 50.6 (13.29) | 50.6 (12.95)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 132 | 126 | 127 | 385
  From 65 to 84 years | 18 | 25 | 23 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 77 | 75 | 237
  Male | 65 | 74 | 75 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 18 | 18 | 58
  Not Hispanic or Latino | 127 | 128 | 132 | 387
  Unknown or Not Reported | 1 | 5 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 5 | 15
  White | 141 | 143 | 141 | 425
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 7 | 9 | 8 | 24
  BULGARIA | 15 | 17 | 21 | 53
  CZECH REPUBLIC | 10 | 10 | 7 | 27
  HUNGARY | 8 | 7 | 9 | 24
  ISRAEL | 3 | 5 | 2 | 10
  MALAYSIA | 1 | 0 | 2 | 3
  POLAND | 39 | 42 | 38 | 119
  RUSSIAN FEDERATION | 10 | 13 | 5 | 28
  SPAIN | 2 | 1 | 4 | 7
  TURKEY | 5 | 4 | 4 | 13
  UKRAINE | 18 | 14 | 18 | 50
  UNITED STATES | 32 | 29 | 32 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response: >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: At Week 24
Population: Full analysis set (FAS) included all participants who were randomized in the study and included in the analyses. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 142 | 146 | 138
Percentage of participants | 35.9 | 63.0 | 60.9

2. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Response of Investigator's Global Assessment (IGA) Psoriasis Score of 0 or 1 and >=2 Grade Reduction From Baseline at Week 24 Among the Participants With >=3 Percent(%) Body Surface Area (BSA)
Description: A psoriasis IGA response was defined as an IGA score of 0 (cleared) or 1 (minimal) and greater than equal to (>=2) grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: At Week 24
Population: Full analysis set included all participants who were randomized in the study and included in the analyses among the participants who had >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 80 | 84 | 81
percentage of participants | 18.8 | 60.7 | 56.8

3. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 90 Response at Week 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 90 response: >=90% improvement in PASI score from baseline.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 80 | 84 | 82
percentage of participants | 12.5 | 47.6 | 54.9

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a participant has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living), each scored from 0 (no difficulty) to 3 (inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Time Frame: Baseline (pre dose Week 0) and Week 24
Population: FAS included all participants who were randomized in the study and included in the analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 150 | 151 | 150
units on a scale | -0.2359 [-0.3200 to -0.1519] | -0.3955 [-0.4787 to -0.3122] | -0.4159 [-0.5006 to -0.3313]

5. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline (pre dose Week 0) and Week 24
Population: FAS included all participants who were randomized in the study and included in the analyses. Missing data were imputed using Multiple Imputation (MI) after applying the Intercurrent Event (ICE) strategies. N (overall number of participants analyzed) included all participants with change data at Week 24 after applying the ICE Strategy and Missing Data Imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 150 | 151 | 150
units on a scale | 3.705 [2.464 to 4.946] | 6.986 [5.758 to 8.213] | 7.027 [5.772 to 8.282]

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 24
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Positive changes from baseline indicate improvement of fatigue. Items were reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: Baseline (pre dose Week 0) and Week 24
Population: FAS included all participants who were randomized in the study and included in the analyses. Missing data were imputed using MI after applying the ICE strategies. N (overall number of participants analyzed) included all participants with change data at Week 24 after applying the ICE Strategy and Missing Data Imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 150 | 151 | 150
units on a scale | 3.9 [2.5 to 5.3] | 7.8 [6.4 to 9.2] | 8.4 [7.0 to 9.9]

7. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Week 24
Description: MDA is a measure that defines a satisfactory state of disease activity that includes 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity on arthritis and psoriasis, physical function and enthesitis). Participants were classified as achieving MDA if they fulfilled 5 of the following 7 criteria at that visit: Tender joint count (68 joints)<=1, Swollen joint count (66 joints) <=1, Psoriasis activity and severity index <=1, Patient's Assessment of Pain <=15 on a 100-unit VAS, Patient's Global Assessment of Disease Activity (arthritis and psoriasis) <=20 on a 100-unit VAS, HAQ-DI score <=0.5, and Tender entheseal points <= 1 (LEI index score <= 1).
Time Frame: At Week 24
Population: Full analysis set included all participants who were randomized in the study and were included in analyses. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 142 | 145 | 137
percentage of participants | 5.6 | 24.8 | 20.4

8. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response at Week 16
Description: as for outcome 1
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 140 | 146 | 139
percentage of participants | 30.7 | 57.5 | 53.2

9. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response at Week 16
Description: ACR 50 response: >=50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 139 | 146 | 140
percentage of participants | 10.1 | 28.8 | 25.0

10. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response at Week 24
Description: as for outcome 9
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: percantage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 142 | 146 | 138
percantage of participants | 12.7 | 32.9 | 33.3

11. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response at Week 24
Description: ACR 70 response: >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Followed by Guselkumab 100 mg | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 141 | 146 | 137
percentage of participants | 2.1 | 17.8 | 19.0

12. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

13. Secondary Outcome: Percentage of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Time Frame: From first administration of study drug (Week 0) up to Week 112
Population: Safety Analysis Set included all participants who received at least one (complete or partial) administration of any study intervention, i.e. the treated population.
Reporting Status: Not Posted, anticipated posting 2027-07

14. Secondary Outcome: Percentage of Participants With Treatment Emergent Related AEs (TERAEs)
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

15. Secondary Outcome: Treatment Emergent AEs Leading to Discontinuation of Study Intervention
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

16. Secondary Outcome: Percentage of Participants With Infections
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

17. Secondary Outcome: Percentage of Participants With Injection-site Reactions
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

18. Secondary Outcome: Percentage of Participants With Infusion Related Reactions
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

19. Secondary Outcome: Number of Participants With Post-baseline Laboratory Abnormalities With Maximum Toxicity Grade Greater Than or Equal to >=3 Based on Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: From first administration of study drug (Week 0) up to Week 112
Reporting Status: Not Posted, anticipated posting 2027-07

20. Secondary Outcome: Serum Guselkumab Concentration Over Time
Description: Serum concentrations of guselkumab over time was reported.
Time Frame: At Weeks 0, 4, 8, 12, 16, 20,and 24
Population: Pharmacokinetics (PK) analysis set all participants who received at least one complete administration of guselkumab and had at least one valid blood sample drawn for PK analysis. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters (mcg/mL)
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 143 | 145
micrograms/milliliters (mcg/mL)
  Week 0 | 0.00 (0.003) | 0.00 (0.004)
  Week 4: number analyzed (Participants) | 140 | 142
  Week 4 | 2.22 (1.162) | 2.32 (1.331)
  Week 8: number analyzed (Participants) | 128 | 129
  Week 8 | 3.23 (1.789) | 3.16 (1.740)
  Week 12: number analyzed (Participants) | 126 | 107
  Week 12 | 1.10 (0.745) | 3.45 (2.038)
  Week 16: number analyzed (Participants) | 112 | 95
  Week 16 | 2.79 (1.436) | 3.58 (2.119)
  Week 20: number analyzed (Participants) | 105 | 89
  Week 20 | 0.90 (0.603) | 3.61 (2.013)
  Week 24: number analyzed (Participants) | 95 | 80
  Week 24 | 2.71 (1.347) | 3.79 (2.288)

21. Secondary Outcome: Number of Participants With Antibodies to Guselkumab
Description: Number of participants with antibodies to guselkumab (ADA) were reported. A validated immunoassay was used to detect ADA.
Time Frame: Baseline (pre dose Week 0) up to Week 24
Population: Immunogenicity analysis set included all participants who received at least one (complete or partial) administration of guselkumab and who had at least 1 sample obtained after their first administration of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 149 | 149
Participants | 6 | 17

ADVERSE EVENTS:
Time Frame: From first administration of study drug (Week 0) up to Week 24
Description: Safety analysis set included all participants who received at least one (complete or partial) administration of any study intervention, that is , the treated population.
Groups:
- Placebo: Participants received placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 24. Participants then received guselkumab 100 mg subcutaneous injections every 4 weeks from Week 24 through to end of study.
- Guselkumab 100 mg q8w: Participants received guselkumab 100 mg subcutaneous injections at Weeks 0 and 4, then every 8 weeks and placebo matched to guselkumab injections at other visits through to end of study.
Arm/Group | Placebo | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/151 | 1/150
Serious Adverse Events (participants affected / at risk) | 6/149 | 4/151 | 2/150
Other Adverse Events (participants affected / at risk) | 18/149 | 24/151 | 16/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Guselkumab 100 mg q8w (N=151) | Guselkumab 100 mg q4w (N=150)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Allergy to Arthropod Sting (Immune system disorders) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myasthenia Gravis (Nervous system disorders) | 0 | 0 | 1
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Guselkumab 100 mg q8w (N=151) | Guselkumab 100 mg q4w (N=150)
Covid-19 (Infections and infestations) | 8 | 8 | 7
Nasopharyngitis (Infections and infestations) | 8 | 9 | 5
Headache (Nervous system disorders) | 3 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the Sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (4):
  • Study Protocol (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04936308/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT04936308/SAP_001.pdf
  • Informed Consent Form: INFORMED CONSENT FORM ADDENDUM (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04936308/ICF_002.pdf
  • Informed Consent Form: MASTER INFORMED CONSENT FORM (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT04936308/ICF_003.pdf